CLINICAL TRIAL: NCT00300898
Title: Radiofrequency Nucleoplasty vs Percutaneous Nucleotomy (Dekompressor) vs Decompression Catheter for the Treatment of Painful Contained Lumbar Disc Herniation: A Prospective Randomized Controlled Study
Brief Title: Radiofrequency Nucleoplasty vs Percutaneous Nucleotomy vs Decompression Catheter in Lumbar Disc Herniation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 8006
Record Dates: First submitted 2006-03-08; First posted 2006-03-10 (Estimated); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Herniated Disc
Keywords: contained lumbar herniated disc; nucleoplasty; percutaneous decompression; Dekompressor; intervertebral electrothermal disc decompression; IDET
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Conservative Treatment

ARMS (4):
- Nucleoplasty (Active Comparator): Procedure/Surgery: Nucleoplasty
  Interventions: Procedure: Nucleoplasty
- Percutaneous decompression (Active Comparator): Procedure/Surgery: Percutaneous decompression
  Interventions: Procedure: Percutaneous decompression
- Electrothermal disc decompression (IDET) (Active Comparator): Procedure/Surgery: Intervertebral electrothermal disc decompression (IDET)
  Interventions: Procedure: Intervertebral electrothermal disc decompression (IDET)
- Behavioral:Conservative treatment (Experimental): Conservative treatment with oral medications, physical therapy, epidural steroid injections
  Interventions: Behavioral: Conservative treatment

INTERVENTIONS:
Procedure: Nucleoplasty
  Arms: Nucleoplasty
Procedure: Percutaneous decompression
  Arms: Percutaneous decompression
Procedure: Intervertebral electrothermal disc decompression (IDET)
  Arms: Electrothermal disc decompression (IDET)
Behavioral: Conservative treatment
  Arms: Behavioral:Conservative treatment

SUMMARY:
The purpose of this study is to learn which of three minimally invasive procedures is the most effective for treatment of contained lumbar disc herniation.

DETAILED DESCRIPTION:
Contained herniation of the lumbar intervertebral disc is a frequent cause of leg and back pain. Over the last decade, there is a tendency to shift from surgical treatment of the intervertebral disc including laminectomy/discectomy to an excess of nonoperative management. Three techniques introduced recently are used as minimally invasive treatments for decompression of contained herniation of the nucleus pulposus. Nucleoplasty uses Coblation® radiofrequency vaporization of nuclear tissue to decompress the intervertebral disc. Catheter disc decompression uses heat from a resistive coil positioned in the area of disc herniation while Dekompressor® uses volume reduction to decrease an intradiscal pressure.

This is a comparison study which investigates if intervertebral electrothermal disc decompression produces better pain relief measured on VAS scale, improvement in functional capacity, return to work and opioid use, than nucleoplasty or percutaneous disc decompression (Dekompressor) of the lumbar intervertebral disc in a prospective randomized controlled study. Patients will be randomized into four treatment groups in equal numbers. The first group will be treated using nucleoplasty, the second will receive Dekompressor® lumbar disc decompression, the third will receive thermal treatment using decompression catheter (Achutherm TM) and the forth will be the control group. The control group will be treated conservatively using medications including gabapentin, a breakthrough opioid (oxycodone 5 mg 1-2 tablets q 4-6 hours as needed), NSAID, epidural steroid injections and physical therapy.

Patients will be followed and assessed at one, three, six, nine and twelve months following the procedure using VAS scores, Oswestry and SF-36 Short Form questionnaires, opioid use and return to work evaluation.

ELIGIBILITY:
Inclusion Criteria:

* History of concordant radicular leg pain unresponsive to conservative treatment for longer than 3 months
* Leg pain must be greater than back pain
* Contained disc herniation as evidenced by MRI
* No evidence of psychological issues by exam or history

Exclusion Criteria:

* A score of greater than 10 on Beck Depression Inventory (BDI)
* Patients with pending workers compensation claim or litigation
* Pregnancy
* Tumor
* Systemic infection or localized infection at the anticipated entry needle site
* Traumatic spinal fracture
* History of coagulopathy
* Unexplained bleeding
* Progressive neurological deficits
* History of opioid abuse or patients currently on long acting opioids
* Patients presenting with moderate or severe lumbar central or lateral canal stenosis, free disc fragments or degenerative disc disease as described on MRI

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2006-07 (Actual); Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
VAS pain evaluation score at baseline, 1, 3, 6, 9, 12 months | baseline 1, 3, 6, 9, 12 months

SECONDARY OUTCOMES:
Oswestry results | baseline 1, 3, 6, 9, 12 months
  Disability Index
Quality of Life SF-36 | baseline 1, 3, 6, 9, 12 months
  SF-36 score at baseline 1, 3, 6, 9, 12 months
Return to work evaluation | 1 month
  Return to work evaluation
Depression score | BASELINE
  Beck Depression Inventory score at pre-treatment visit
Opioid use | 1, 3, 6, 9, 12 months
  Opioid use

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Kapural, MD, OhD, Principal Investigator — Cleveland Clinic Foundation, Pain Management Department

IPD SHARING:
Plan to Share IPD: No